CLINICAL TRIAL: NCT00405821
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Acyclovir Prophylaxis Versus Placebo Among HIV-1/HSV-2 Co-Infected Individuals in Uganda
Brief Title: Acyclovir to Treat Patients Co-infected With HIV and Herpes Viruses in Uganda
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Washington (Other); Johns Hopkins University (Other); Translational Genomics Research Institute (Other)
Responsible Party: Principal Investigator, Steven Reynolds, Scientific Director NIH-Uganda ICER, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999907032; 07-I-N032 (Other: NIAID Intramural IRB)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-08

CONDITIONS: HIV Infections; Herpes Genitalis
Keywords: AIDS; HIV Disease Progression; Quality of Life; HIV Viral Load; Genital Ulcers; HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections; Herpes Genitalis; Acquired Immunodeficiency Syndrome | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acyclovir 400mg tablet twice daily (Active Comparator)
  Interventions: Drug: Acyclovir
- Placebo tablet twice daily (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acyclovir — 400mg twice daily for 24 months
  Arms: Acyclovir 400mg tablet twice daily
Drug: Placebo — Placebo tablet twice daily for 24 months
  Arms: Placebo tablet twice daily

SUMMARY:
This study will determine whether acyclovir, a medicine used to treat herpes simplex virus 2 (HSV-2), can slow down the progression (worsening) of HIV disease in people with both HIV and HSV-2 infections. HSV-2 increases the amount of HIV virus in the blood of infected people and may make HIV progress faster. The study will evaluate:

"Whether people who take acyclovir can avoid antiretroviral treatment until later in their lives

"Whether people who take acyclovir get fewer genital ulcers

"How well people are able to take acyclovir and any side effects they experience from it

"Differences in the amount of HIV virus in the blood of patients who are and are not taking acyclovir, and how HIV/AIDS is different in these patients.

People 18 years of age and older living in the Rakai district of Uganda who are infected with both HIV (early stage disease) and HSV-2 may be eligible for this study. Participants are randomly assigned to take the study drug, acyclovir, or a placebo (look-alike pill with no active ingredient) daily for 2 years. During this time, they visit the clinic once a month for a routine physical examination. Patients who develop genital ulcers or complications of HIV are treated for the problem, and patients whose HIV disease progresses, requiring them to begin antiretroviral therapy, are treated accordingly.

DETAILED DESCRIPTION:
Interventions that slow HIV-1 disease progression among persons with CD4+ counts above 250 cells/microliter could postpone the need for antiretroviral therapy (ART) and prolong life-expectancy for HIV-infected persons. Herpes simplex virus type 2 (HSV-2) has been shown to up-regulate HIV-1 replication at the cellular level. (1) This finding has been supported by clinical evidence that individuals who are HSV-2 seropositive at the time of HIV-1 seroconversion had higher HIV viral loads at 5 and 15 months post-seroconversion. (2) Earlier studies during the era of zidovudine (Retrovir) monotherapy showed a survival advantage when acyclovir (ACV, Zovirax) was added to the treatment of patients with HIV. (3) Acyclovir prophylaxis has been shown to decrease herpes simplex virus infections and varicella-zoster virus infections among HIV infected patients in a meta-analysis of randomized trials from North America and Europe. This analysis also found a reduced risk of mortality among patients treated with acyclovir. The potential of acyclovir to slow HIV-1 disease progression has not been assessed in a randomized trial in Africa where high rates of HSV-2 infection have been observed among HIV-1 infected individuals. This study proposes to assess the benefits of acyclovir prophylaxis among HIV-1 infected individuals dually infected with HSV-2 who are not on ART through a randomized double-blind placebo controlled trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Documentation of HIV-1 infection, by either two positive ELISAs or two discrepant ELISAs with a confirmatory positive Western Blot
  2. Documentation of prior HSV-2 infection by Focus Kalon ELISA
  3. Absolute CD4+ T-cell count of greater than or equal to 300 and less than or equal to 400 cells/microliter within 30 days prior to randomization
  4. All participants must be receiving Cotrimoxazole prophylaxis as part of standard care unless contraindicated
  5. Age at least 18 years and above
  6. Laboratory values (within 30 days prior to randomization)

     1. Aspartate transaminase (AST) no more than five times the upper limit of normal (ULN)
     2. Total bilirubin no more than 2 times ULN
     3. Creatinine no more than 2.0 mg/dL
     4. Platelet count at least 50 000/microliter
     5. Hemoglobin at least 8g/dL
  7. Written informed consent

EXCLUSION CRITERIA:

1. Concurrent malignancy or any other disease state requiring cytotoxic chemotherapy
2. Symptomatic for significant HIV-related illnesses (WHO stage III or IV), such as opportunistic infections and malignancies other than mucocutaneous Kaposi's sarcoma. A history of AIDS defining opportunistic infections other than mucocutaneous Kaposi's sarcoma or candida or treated tuberculosis
3. Active HSV-2 disease as suggested by painful genital ulcer disease at time of screening or enrollment
4. Current use of antiretroviral medications or Preventing Mother-to-Child Transmission (PMTCT) use of antiretrovirals within the previous 6 months
5. Significant cardiac, pulmonary, kidney, rheumatologic, gastrointestinal, or CNS disease as detectable on routine medical history, physical examination, or screening laboratory studies.
6. Psychiatric illness that, in the opinion of the PI, might interfere with the study compliance.
7. Active substance abuse or history of prior substance abuse that may interfere with protocol compliance or patient safety.
8. CD4+ count less than 300 or more than 400 cells/microliter.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2006-11; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Rakai Health Sciences Program, Uganda Virus Research Institute, Kalisizo, Rakai District, Uganda

REFERENCES:
- [Background] Moriuchi M, Moriuchi H, Williams R, Straus SE. Herpes simplex virus infection induces replication of human immunodeficiency virus type 1. Virology. 2000 Dec 20;278(2):534-40. doi: 10.1006/viro.2000.0667. PMID 11118375
- [Background] Serwadda D, Gray RH, Sewankambo NK, Wabwire-Mangen F, Chen MZ, Quinn TC, Lutalo T, Kiwanuka N, Kigozi G, Nalugoda F, Meehan MP, Ashley Morrow R, Wawer MJ. Human immunodeficiency virus acquisition associated with genital ulcer disease and herpes simplex virus type 2 infection: a nested case-control study in Rakai, Uganda. J Infect Dis. 2003 Nov 15;188(10):1492-7. doi: 10.1086/379333. Epub 2003 Oct 28. PMID 14624374
- [Background] Stein DS, Graham NM, Park LP, Hoover DR, Phair JP, Detels R, Ho M, Saah AJ. The effect of the interaction of acyclovir with zidovudine on progression to AIDS and survival. Analysis of data in the Multicenter AIDS Cohort Study. Ann Intern Med. 1994 Jul 15;121(2):100-8. doi: 10.7326/0003-4819-121-2-199407150-00004. PMID 8017721
- [Derived] Redd AD, Newell K, Patel EU, Nalugoda F, Ssebbowa P, Kalibbala S, Frank MA, Tobian AA, Gray RH, Quinn TC, Serwadda D, Reynolds SJ. Decreased monocyte activation with daily acyclovir use in HIV-1/HSV-2 coinfected women. Sex Transm Infect. 2015 Nov;91(7):485-8. doi: 10.1136/sextrans-2014-051867. Epub 2015 Apr 22. PMID 25904747
- [Derived] Reynolds SJ, Makumbi F, Newell K, Kiwanuka N, Ssebbowa P, Mondo G, Boaz I, Wawer MJ, Gray RH, Serwadda D, Quinn TC. Effect of daily aciclovir on HIV disease progression in individuals in Rakai, Uganda, co-infected with HIV-1 and herpes simplex virus type 2: a randomised, double-blind placebo-controlled trial. Lancet Infect Dis. 2012 Jun;12(6):441-8. doi: 10.1016/S1473-3099(12)70037-3. Epub 2012 Mar 19. PMID 22433279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 440 HIV+ subjects recruited in rural Rakai, Uganda within the Rakai Health Sciences Program mobile medical clinic during May 2007 thru November 2008
Pre-assignment Details: All subjects were randomized to study arm, and initiated study treatment at the time of enrollment.
Period: Overall Study
Arm/Group | Acyclovir 400mg Tablet Twice Daily | Placebo Tablet Twice Daily
Started | 220 | 220
Completed | 198 | 198
Not Completed | 22 | 22
Not completed — Death | 5 | 7
Not completed — Lost to Follow-up | 7 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — initiated ART | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acyclovir 400mg Tablet Twice Daily | Placebo Tablet Twice Daily | Total
Number analyzed (Participants) | 220 | 220 | 440
Age, Customized [Number; unit: participants]
  20-29 years | 46 | 44 | 90
  30-39 years | 94 | 93 | 187
  40-49 years | 54 | 53 | 107
  50+ years | 26 | 30 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 161 | 311
  Male | 70 | 59 | 129

OUTCOME MEASURES:

1. Primary Outcome: Progression to AIDS (CD4+ Less Than 250 Cells/Microliter or World Health Org Stage IV dx, Excluding Esophageal Candidiasis)
Description: Evaluate the effect of acyclovir prophylaxis vs placebo among HIV-1/HSV-2 co-infected individuals on the progression to AIDS (CD4+ less than 250 cells/microliter or World Health Org stage IV disease, excluding esophageal candidiasis)
Time Frame: 2 years
Population: Intention to treat analysis of all subjects randomized on the trial meeting the primary endpoint
Measure: Number; unit: participants
Arm/Group | Acyclovir 400mg Tablet Twice Daily | Placebo Tablet Twice Daily
Number analyzed (Participants) | 220 | 220
participants | 95 | 110
Statistical Analysis 1: Comparison: Acyclovir 400mg Tablet Twice Daily vs Placebo Tablet Twice Daily; Intent-to-treat analysis used Cox proportional hazards (CPH) models, adjusting for baseline log10 viral load (VL), CD4 cell count, gender and age to assess the risk of disease progression; Test type: Superiority or Other; p < 0.05, Regression, Cox — P-value was adjusted to include multiple looks at data including an interim efficacy review at 50% and 75% accrual of person-years on study; adjusted for baseline log10 viral load, baseline CD4 count, gender, and age; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.58 to 0.99]

2. Secondary Outcome: Difference in Number of Episodes of Genital Ulcer Disease Between Arms
Description: We calculated incidence rate for each treatment arm for episodes of genital ulcer disease, and incidence rate ratio.
Time Frame: 2 years
Population: We conducted monthly clinical assessment for GUD on all randomized subjects during their entire follow-up period on this trial. The number of episodes of GUD is shown below.
Measure: Number; unit: episodes
Arm/Group | Acyclovir 400mg Tablet Twice Daily | Placebo Tablet Twice Daily
Number analyzed (Participants) | 220 | 220
episodes | 27 | 47
Statistical Analysis 1: Comparison: Acyclovir 400mg Tablet Twice Daily vs Placebo Tablet Twice Daily; Null hypothesis is no difference by treatment arm in rate of GUD; Test type: Superiority or Other; p < 0.05, rate ratio with 95% CI — we included multiple GUD events per subject in the estimate of GUD incidence; Risk Ratio (RR) = 0.31, 95% CI 2-sided [0.19 to 0.48]

3. Secondary Outcome: HIV-1 Viral Load Difference Between Arms
Description: We measured mean annual rate of change in log10 viral load (copies/mL) for each group. We assessed difference in annual rate of change in log10 viral load (copies/mL) between groups.
Time Frame: baseline, 6 months, 12 months, 18 months, 24 months
Population: We measured viral load at baseline and at 6 monthly follow-up visits during 24 months of follow-up for all subjects randomized on this study.
Measure: Mean (95% Confidence Interval); unit: log10 (copies/mL)
Arm/Group | Acyclovir 400mg Tablet Twice Daily | Placebo Tablet Twice Daily
Number analyzed (Participants) | 220 | 220
log10 (copies/mL) | -0.061 [-0.250 to 0.129] | 0.402 [0.212 to 0.592]
Statistical Analysis 1: Comparison: Acyclovir 400mg Tablet Twice Daily vs Placebo Tablet Twice Daily; Null hypothesis is no difference in annual rate of change in log10 viral load by arm; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.463, 95% CI 2-sided [-0.731 to -0.194]

4. Secondary Outcome: Toxicity of Acyclovir
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Adherence to Acyclovir
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Virologic and Immunologic Responses to ART in Those Who Progress to CD+4 Less Than 250cells/mL
Time Frame: 6 months and 12 moths post ART initiation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: maximum follow-up time on this study ranged from 24 months to 41 months depending on time of enrollment.
Arm/Group | Acyclovir 400mg Tablet Twice Daily | Placebo Tablet Twice Daily
Serious Adverse Events (participants affected / at risk) | 75/220 | 85/220
Other Adverse Events (participants affected / at risk) | 219/220 | 218/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir 400mg Tablet Twice Daily (N=220) | Placebo Tablet Twice Daily (N=220)
TB Adenitis (Infections and infestations) | 1 (1) | 1 (1)
Malaria (Infections and infestations) | 26 (29) | 24 (34)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (9) | 13 (16)
Dehydration (General disorders) | 1 (1) | 0 (0)
Febrile Illness, unspecified (General disorders) | 5 (5) | 5 (6)
skin infection, unspecified (Infections and infestations) | 1 (1) | 1 (1)
wound, unspecified (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
EENT infection, unspecified (Infections and infestations) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Bacterial pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pulmonary Tuberculosis (Infections and infestations) | 13 (13) | 13 (14)
Extra-pulmonary tuberculosis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory complaint, unspecified (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cryptococcal meningitis (Infections and infestations) | 0 (0) | 1 (1)
Esophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Peptic ulcer disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain, unspecified (Gastrointestinal disorders) | 1 (1) | 3 (3)
Trauma to chest (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic inflammatory disease (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Genito-urinary disease (GUD) (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 30 (37) | 41 (52)
Pregnancy complication, unspecified (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 2 (2)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir 400mg Tablet Twice Daily (N=220) | Placebo Tablet Twice Daily (N=220)
Malaria (Infections and infestations) | 107 (211) | 105 (204)
Lymphadenopathy (General disorders) | 25 (30) | 36 (47)
Decreased appetite (General disorders) | 30 (35) | 29 (33)
General complaint, unspecified (General disorders) | 190 (791) | 187 (810)
Herpes zoster (Skin and subcutaneous tissue disorders) | 4 (4) | 18 (18)
fungal skin infection (Infections and infestations) | 64 (102) | 46 (70)
angular chelitis (Infections and infestations) | 21 (23) | 34 (45)
Papulo-pruritic eruption (PPE) (Skin and subcutaneous tissue disorders) | 15 (21) | 22 (27)
Darkening nails (Skin and subcutaneous tissue disorders) | 31 (32) | 32 (32)
Rash, unspecified (Skin and subcutaneous tissue disorders) | 118 (227) | 119 (201)
Skin complaint, unspecified (Skin and subcutaneous tissue disorders) | 123 (213) | 122 (212)
Rhinitis (Infections and infestations) | 20 (20) | 18 (20)
Conjunctivitis (Infections and infestations) | 29 (34) | 32 (40)
Allergic conjunctivitis (Eye disorders) | 33 (41) | 21 (29)
Hearing Loss (Ear and labyrinth disorders) | 14 (16) | 15 (16)
General complaint, unspecified (General disorders) | 115 (217) | 123 (252)
Palpitations (Cardiac disorders) | 32 (41) | 41 (58)
Upper respiratory tract infection (Infections and infestations) | 212 (1242) | 212 (1226)
Respiratory complaint, unspecified (Respiratory, thoracic and mediastinal disorders) | 98 (152) | 82 (132)
HIV neuritis (Nervous system disorders) | 36 (45) | 22 (24)
post-herpetic neuralgia (Nervous system disorders) | 7 (8) | 15 (20)
Nervous system, other complaint (Nervous system disorders) | 55 (76) | 46 (68)
Oral candidiasis (Infections and infestations) | 15 (26) | 23 (40)
Peptic ulcer disease (Gastrointestinal disorders) | 63 (124) | 60 (115)
Intestinal helminthiasis (Infections and infestations) | 12 (12) | 20 (25)
Gastroenteritis (Infections and infestations) | 41 (55) | 33 (55)
Gastritis (Gastrointestinal disorders) | 27 (31) | 33 (42)
Gastrointestinal, other complaint (Gastrointestinal disorders) | 168 (415) | 157 (488)
Arthritis (Musculoskeletal and connective tissue disorders) | 19 (23) | 15 (18)
Traumatic injury (Injury, poisoning and procedural complications) | 16 (18) | 16 (16)
Musculoskeletal joint pain, unspecified (Musculoskeletal and connective tissue disorders) | 165 (470) | 162 (472)
Pelvic inflammatory disease (Reproductive system and breast disorders) | 21 (22) | 21 (24)
Gonorrhea (Infections and infestations) | 14 (20) | 12 (14)
Genito-urinary disease (GUD) (Infections and infestations) | 39 (52) | 77 (131)
Vaginal candidiasis (Infections and infestations) | 80 (134) | 79 (159)
Urinary Tract Infection (Infections and infestations) | 36 (48) | 39 (55)
Vaginal discharge (Reproductive system and breast disorders) | 10 (10) | 14 (16)
Genitourinary, other complaint (Reproductive system and breast disorders) | 131 (280) | 140 (356)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes